CLINICAL TRIAL: NCT00334633
Title: Tinidazole for the Treatment of Bacterial Vaginosis
Brief Title: Treatment of Bacterial Vaginosis (BV) With Tinidazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Jane Schwebke, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F040329003; R01AI058033 (NIH)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; tinidazole
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Tinidazole; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- control (Active Comparator): metronidazole 500 BID for 7 days
  Interventions: Drug: tinidazole, metronidazole
- tinidazole 500 (Active Comparator): tinidazole 500 BID for 7 days
  Interventions: Drug: tinidazole, metronidazole
- tinidazole 1 gm (Active Comparator): tinidazole 1 gm BID for 7 days
  Interventions: Drug: tinidazole, metronidazole

INTERVENTIONS:
Drug: tinidazole, metronidazole — Tinidazole 500 mg bid; Tinidazole 1mg bid; Metronidazole 500mg bid
  Other Names: Tindamax, Flagyl

SUMMARY:
We are trying to determine if treatment of bacterial vaginosis with tinidazole is better than treatment with metronidazole

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is the most prevalent cause of symptomatic vaginal discharge in the U.S. and has been associated with complications including preterm delivery of infants, pelvic inflammatory disease (PID), urinary tract infections (UTI) and acquisition/transmission of sexually transmitted diseases (STDs) including human immunodeficiency virus (HIV). Control of BV has been advocated as a means of decreasing the prevalence of these complications. However, the etiology of BV remains unknown and the current treatment regimens are inadequate in terms of initial cure and recurrence rates. Although not currently licensed in the U.S., tinidazole is an antimicrobial related to metronidazole which has shown promise for the treatment of BV in European studies and is widely used worldwide for the treatment of trichomoniasis including infections which are resistant to metronidazole. We hypothesize that qualities of tinidazole such as its longer half-life and its seemingly superior side effect profile as compared to oral metronidazole will result in its being a more efficacious drug for the treatment of BV than the currently available options.

The specific aims of this project are:

1. To compare the efficacy of two different doses of tinidazole with oral metronidazole for the initial treatment of symptomatic BV as well as short-term recurrence rates
2. To compare the side effect profiles of tinidazole versus metronidazole in the treatment of BV
3. To compare drug levels of tinidazole and metronidazole in the vaginal secretions and correlate with microbiologic cure of BV as well as rates of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Women be at least 18 years of age
* Have symptoms of vaginal odor and or/discharge
* Meet the clinical (Amsel) criteria for BV
* Willing to participate in research

Exclusion Criteria:

* Presence of another vaginal infection or STD
* Allergy to metronidazole
* Pregnant or nursing
* Use of oral or intravaginal antibiotics within the past 2 weeks
* HIV or other chronic disease
* Inability to keep return appointments

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 593 (Actual)
Dates: Start 2004-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Schwebke, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Jefferson County Department of Health STD Clinic, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: women attending a sexually transmitted disease (STD) clinic with symptomatic bacterial vaginosis (BV)
Groups:
- Metronidazole: metronidazole 500 twice a day (BID) for 7 days; 197 participants
- Tinidazole 500 mg: tinidazole 500 BID for 7 days; 200 particpants
- Tinidazole 1 gm: tinidazole 1 gm BID for 7 days; 196 particpants
Period: Overall Study
Arm/Group | Metronidazole | Tinidazole 500 mg | Tinidazole 1 gm
Started | 197 | 200 | 196
Completed | 117 | 118 | 114
Not Completed | 80 | 82 | 82

BASELINE CHARACTERISTICS:
Groups:
- Metronidazole: metronidazole 500 BID for 7 days; 197 participants
- Total: Total of all reporting groups
Arm/Group | Metronidazole | Tinidazole 500 mg | Tinidazole 1 gm | Total
Number analyzed (Participants) | 197 | 200 | 196 | 593
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 197 | 200 | 196 | 593
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6.2) | 28.3 (6.6) | 28.5 (6.8) | 28.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 200 | 196 | 593
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 197 | 200 | 196 | 593

OUTCOME MEASURES:

1. Primary Outcome: Cure of Bacterial Vaginosis
Description: resolution of Amsel criteria for bacterial vaginosis
Time Frame: one month
Population: ITT
Measure: Number; unit: participants
Arm/Group | Metronidazole | Tinidazole 500 mg | Tinidazole 1 gm
Number analyzed (Participants) | 117 | 118 | 114
participants | 75 | 73 | 77

2. Secondary Outcome: Recurrence of BV
Time Frame: baseline to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Tinidazole 500 | Tinidazole 1 gm
Number analyzed (Participants) | 117 | 114 | 118
Participants | 42 | 45 | 37

ADVERSE EVENTS:
Arm/Group | Metronidazole | Tinidazole 500 mg | Tinidazole 1 gm
Serious Adverse Events (participants affected / at risk) | 0/197 | 0/200 | 0/196
Other Adverse Events (participants affected / at risk) | 87/197 | 109/200 | 145/196
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Metronidazole (N=197) | Tinidazole 500 mg (N=200) | Tinidazole 1 gm (N=196)
vaginal candidiasis (Infections and infestations) | 32/126 (32) | 33/161 (33) | 27 (27)
gastrointestinal (Gastrointestinal disorders) | 39/126 (39) | 54/161 (54) | 91 (91)
headache (Nervous system disorders) | 16/126 (16) | 22/161 (22) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No